CLINICAL TRIAL: NCT05263206
Title: Master Protocol of Two Randomized, Double Blind, Placebo-controlled, Multi-center, Parallel Group Studies to Evaluate the Efficacy and Safety of Dupilumab in Adult Patients With Chronic Pruritus of Unknown Origin (CPUO)
Brief Title: Efficacy and Safety of Subcutaneous Dupilumab for the Treatment of Adult Participants With Chronic Pruritus of Unknown Origin (CPUO) (LIBERTY-CPUO-CHIC)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EFC16973; U1111-1253-9888 (Registry Identifier: ICTRP); 2023-508879-36-00 (Registry Identifier: CTIS); 2023-508879-36 (Registry Identifier: CTIS); 2021-004315-76 (EudraCT Number)
Record Dates: First submitted 2022-02-22; First posted 2022-03-02 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Pruritus
MeSH Terms: conditions — Pruritus | interventions — dupilumab; fexofenadine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dupilumab (Experimental): Loading dose administered subcutaneous (SC), followed by SC once every 2 weeks (Q2W) on top of non-sedative antihistamine and moisturizer
  Interventions: Drug: Dupilumab; Drug: Fexofenadine (loratadine if not available)
- Placebo (Placebo Comparator): Loading dose administered SC, followed by SC Q2W on top of non-sedative antihistamine and moisturizer
  Interventions: Drug: Placebo; Drug: Fexofenadine (loratadine if not available)

INTERVENTIONS:
Drug: Dupilumab — Injection solution subcutaneous
  Arms: Dupilumab
Drug: Placebo — Injection solution SC
  Arms: Placebo
Drug: Fexofenadine (loratadine if not available) — Tablet or capsule Oral

SUMMARY:
The main objective of the study is to assess efficacy and safety of dupilumab given up to 24 weeks in adults with CPUO.

This is a master protocol which includes 2 parallel-treatment, double-blind, 2- arm Phase 3 staggered studies of similar design (Study A and Study B) in male and female participants aged 18 to 90 years with CPUO. Study B design was to be adapted based on the results of Study A.

For both Study A and B, after an up-to-4-week screening period, participants with severe pruritus (worst-itch numerical rating scale [WI-NRS ≥7) will enter a 4-week run-in period and will be treated with a non-sedative antihistamine and an emollient (moisturizer). Participants with severe pruritus (WI-NRS ≥7) at baseline will be randomized (1:1) to be treated for 24 weeks with either dupilumab or matching placebo in addition to their non-sedative antihistamine and emollient regimen. The treatment period for both study A and B will be followed by a 12-week follow-up period.

DETAILED DESCRIPTION:
Study duration per participant will be up to 44 weeks for both Study A and Study B.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be 18 (or the legal age of consent in the jurisdiction in which the study is taking place) to 90 years of age inclusive, at the time of signing the informed consent.
* Participants with chronic pruritus for at least 6 months before the screening visit.
* Chronic pruritus considered of unknown origin as assessed by the investigator at baseline (excluding chronic pruritus secondary to dermatological or systemic conditions, of neuropathic or psychogenic origin or secondary to drugs).
* Chronic pruritus must affect at least 2 of the following body areas: legs, arms, or trunk.
* History of insufficient control of the chronic pruritus with prior treatment.
* Participants should receive optimal treatment for concomitant conditions that could impact pruritus (eg, diabetes, iron deficiency).
* Participants must have a history of severe itch and a worst itch score of ≥7 at screening on the WI-NRS (score scale ranges from 0 to 10; higher score indicates worse itch) and Patient Global Impression of Severity (PGIS) of pruritus scored "severe" at screening.
* Participants must have an average worst itch score of ≥7 in the 7 days prior to run-in visit and in the 7 days prior to Day 1 on the WI-NRS.
* Participants scored "severe" in the PGIS of pruritus on Day 1.

Exclusion Criteria:

Participants are excluded from the study if any of the following criteria apply:

* Severe concomitant illness(es) that, in the Investigator's judgment, would adversely affect the patient's participation in the study.
* Patients with active tuberculosis or non-tuberculous mycobacterial infection, or a history of incompletely treated tuberculosis, unless it is well documented by a specialist that the participant has been adequately treated and can now start treatment with a biologic agent.
* Diagnosed with, suspected of, or at high risk of endoparasitic infection, and/or use of antiparasitic drug within 2 weeks before the screening visit.
* HIV infection.
* Severe renal failure (dialysis).
* Active chronic or acute infection requiring treatment with systemic antibiotics, antivirals, or antifungals within 2 weeks before the run-in visit.
* Known or suspected immunodeficiency.
* Active malignancy or history of malignancy within 5 years before the baseline visit, except completely treated in situ carcinoma of the cervix and completely treated and resolved non metastatic squamous or basal cell carcinoma of the skin.
* History of hypersensitivity or intolerance to non-sedative antihistamines.
* Participation in prior dupilumab clinical study or have been treated with commercially available dupilumab.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 284 (Estimated)
Dates: Start 2022-02-15 (Actual); Primary Completion 2027-06-02 (Estimated); Study Completion 2027-08-25 (Estimated)

PRIMARY OUTCOMES:
Study A: Proportion of participants with improvement (reduction) in weekly average of daily worst-itch numerical rating scale (WI-NRS) by ≥4 from baseline to Week 24 | Baseline to Week 24
  WI-NRS is a patient reported outcome (PRO) comprised of a single item rated on a scale from 0 ("No itch") to 10 ("Worst imaginable itch").
Study B: Proportion of participants with improvement (reduction) in weekly average of daily WI-NRS by ≥4 from baseline to Week 12 | Baseline to Week 12
  WI-NRS is a PRO comprised of a single item rated on a scale from 0 ("No itch") to 10 ("Worst imaginable itch").

SECONDARY OUTCOMES:
Study A; Proportion of participants with improvement (reduction) in weekly average of daily WI-NRS by ≥4 from baseline to Week 12 | Baseline to Week 12
  WI-NRS is a PRO comprised of a single item rated on a scale from 0 ("No itch") to 10 ("Worst imaginable itch").
Study A: Proportion of participants who scored "none" or "mild" in Patient Global Impression of Severity (PGIS) of pruritus at Week 24 | Week 24
  The PGIS of pruritus is a one-item categorical scale that asks participants to provide the overall self-assessment of their pruritus severity on a 4-point scale for the past week. Response choices are: "None", "Mild", "Moderate", "Severe".
Study A: Proportion of participants with improvement (reduction) in weekly average of daily WI-NRS by ≥4 from baseline over time until Week 24 | Baseline to Week 24
  WI-NRS is a PRO comprised of a single item rated on a scale from 0 ("No itch") to 10 ("Worst imaginable itch").
Study A: Time to first response of WI-NRS ≥4 points reduction from baseline by Week 24 | Baseline to Week 24
  WI-NRS is a PRO comprised of a single item rated on a scale from 0 ("No itch") to 10 ("Worst imaginable itch").
Study A: Absolute change from baseline in weekly average of daily WI-NRS at Week 24 | Baseline to Week 24
  WI-NRS is a PRO comprised of a single item rated on a scale from 0 ("No itch") to 10 ("Worst imaginable itch").
Study A: Percent change from baseline in weekly average of daily WI-NRS at Week 24 | Baseline to Week 24
  WI-NRS is a PRO comprised of a single item rated on a scale from 0 ("No itch") to 10 ("Worst imaginable itch").
Study A: Proportion of participants who scored "none" or "mild" in PGIS of pruritus at Week 12 | Week 12
  The PGIS of pruritus is a one-item categorical scale that asks participants to provide the overall self-assessment of their pruritus severity on a 4-point scale for the past week. Response choices are: "None", "Mild", "Moderate", "Severe".
Study A: Absolute change from baseline in weekly average of daily WI-NRS at Week 12 | Baseline to Week 12
  WI-NRS is a PRO comprised of a single item rated on a scale from 0 ("No itch") to 10 ("Worst imaginable itch").
Study A: Percent change from baseline in weekly average of daily WI-NRS at Week 12 | Baseline to Week 12
  WI-NRS is a PRO comprised of a single item rated on a scale from 0 ("No itch") to 10 ("Worst imaginable itch").
Study A: Absolute change from baseline in weekly average of daily sleep disturbance numerical rating scale (NRS) at Week 24 | Baseline to Week 24
  The sleep disturbance NRS is to be used by the participants to report the degree of their sleep loss related to itch over the past 24 hours. Participants will rate their sleep disturbance from 0 ('no sleep loss related to itch') to 10 ('I cannot sleep at all due to itch') once daily in the morning.
Study A: Percent change from baseline in weekly average of daily sleep disturbance NRS at Week 24 | Baseline to Week 24
  The sleep disturbance NRS is to be used by the participants to report the degree of their sleep loss related to itch over the past 24 hours. Participants will rate their sleep disturbance from 0 ('no sleep loss related to itch') to 10 ('I cannot sleep at all due to itch') once daily in the morning.
Study A: Change from baseline in Dermatology Life Quality Index (DLQI) score at Week 24 | Baseline to Week 24
  The DLQI is a validated 10-item questionnaire to measure dermatology-specific quality of life (QoL) in adult patients. Overall scoring ranges from 0 to 30, with a higher score indicating a poorer QoL.
Study A: Change from baseline in the Itchy quality of life (ItchyQoL) score at Week 24 | Baseline to Week 24
  ItchyQoL is a pruritus-specific QoL instrument that measures specifically disease burden in pruritus patients.
Study A: Change from baseline in Hospital Anxiety and Depression Scale (HADS) total score at Week 24 | Baseline to Week 24
  The HADS is a validated questionnaire for screening anxiety and depression in non-psychiatric populations. The total score ranges from 0 to 42. 0 to 7= normal; 8 to 10= borderline abnormal; 11 to 21= abnormal.
Study A: Absolute change from baseline in weekly average of daily sleep disturbance NRS at Week 12 | Baseline to Week 12
  The sleep disturbance NRS is to be used by the participants to report the degree of their sleep loss related to itch over the past 24 hours. Participants will rate their sleep disturbance from 0 ('no sleep loss related to itch') to 10 ('I cannot sleep at all due to itch') once daily in the morning.
Study A: Percent change from baseline in weekly average of daily sleep disturbance NRS at Week 12 | Baseline to Week 12
  The sleep disturbance NRS is to be used by the participants to report the degree of their sleep loss related to itch over the past 24 hours. Participants will rate their sleep disturbance from 0 ('no sleep loss related to itch') to 10 ('I cannot sleep at all due to itch') once daily in the morning.
Study A: Change from baseline in DLQI score at Week 12 | Baseline to Week 12
  The DLQI is a validated 10-item questionnaire to measure dermatology-specific quality of life (QoL) in adult patients. Overall scoring ranges from 0 to 30, with a higher score indicating a poorer QoL.
Study A: Change from baseline in the ItchyQoL score at Week 12 | Baseline to Week 12
  ItchyQoL is a pruritus-specific QoL instrument that measures specifically disease burden in pruritus patients. It is a 22-item instrument that measures the degree to which pruritus affects quality-of-life for the past week. The overall score is the average of the 22 items ranging from 1 to 5. A higher score corresponds to a more adverse impact on QoL.
Study A: Change from baseline in HADS total score at Week 12 | Baseline to Week 12
  The HADS is a validated questionnaire for screening anxiety and depression in non-psychiatric populations. The total score ranges from 0 to 42. 0 to 7= normal; 8 to 10= borderline abnormal; 11 to 21= abnormal.
Study A: Percentage of participants experiencing treatment-emergent adverse events (TEAEs) or serious adverse events (SAEs) from baseline through end of study (EOS) | Baseline to Week 36
  Percentage of participants experiencing TEAEs or SAEs from baseline through EOS
Study A: Incidence of treatment-emergent antidrug antibodies (ADA) against dupilumab | Baseline to Week 36
  Incidence of treatment-emergent ADA against dupilumab
Study B: Proportion of participants who scored "none" or "mild" in PGIS of pruritus at Week 24 | Week 24
  The PGIS of pruritus is a one-item categorical scale that asks participants to provide the overall self-assessment of their pruritus severity on a 4-point scale for the past week. Response choices are: "None", "Mild", "Moderate", "Severe".
Study B: Proportion of participants who scored "none" or "mild" in PGIS of pruritus at Week 12 | Week 12
  The PGIS of pruritus is a one-item categorical scale that asks participants to provide the overall self-assessment of their pruritus severity on a 4-point scale for the past week. Response choices are: "None", "Mild", "Moderate", "Severe".
Study B: Absolute change from baseline in weekly average of daily WI-NRS at Week 12 | Baseline to Week 12
  WI-NRS is a PRO comprised of a single item rated on a scale from 0 ("No itch") to 10 ("Worst imaginable itch").
Study B: Percent change from baseline in weekly average of daily WI-NRS at Week 12 | Baseline to Week 12
  WI-NRS is a PRO comprised of a single item rated on a scale from 0 ("No itch") to 10 ("Worst imaginable itch").
Study B: Absolute change from baseline in weekly average of daily WI-NRS at Week 24 | Baseline to Week 24
  WI-NRS is a PRO comprised of a single item rated on a scale from 0 ("No itch") to 10 ("Worst imaginable itch").
Study B: Percentage change from baseline in weekly average of daily WI-NRS at Week 24 | Baseline to Week 24
  WI-NRS is a PRO comprised of a single item rated on a scale from 0 ("No itch") to 10 ("Worst imaginable itch").
Study B: Proportion of participants with improvement (reduction) in weekly average of daily WI-NRS by ≥4 from baseline, sustained from Week 19 through Week 24 | Baseline to Week 19 through Week 24
  WI-NRS is a PRO comprised of a single item rated on a scale from 0 ("No itch") to 10 ("Worst imaginable itch").
Study B: Proportion of participants with improvement (reduction) in weekly average of daily WI-NRS by ≥5 from baseline to Week 24 | Baseline to Week 24
  WI-NRS is a PRO comprised of a single item rated on a scale from 0 ("No itch") to 10 ("Worst imaginable itch").
Study B: Proportion of participants with improvement (reduction) in weekly average of daily WI-NRS by ≥4 from baseline to Week 24 | Baseline to Week 24
  WI-NRS is a PRO comprised of a single item rated on a scale from 0 ("No itch") to 10 ("Worst imaginable itch").
Study B: Proportion of participants with weekly average of daily WI-NRS <2 at Week 24 | Week 24
  WI-NRS is a PRO comprised of a single item rated on a scale from 0 ("No itch") to 10 ("Worst imaginable itch").
Study B: Time to first response of WI-NRS ≥4 points reduction from baseline by Week 24 | Baseline to Week 24
  WI-NRS is a PRO comprised of a single item rated on a scale from 0 ("No itch") to 10 ("Worst imaginable itch").
Study B: Proportion of participants with improvement (reduction) in weekly average of daily WI-NRS by ≥5 from baseline to Week 12 | Baseline to Week 12
  WI-NRS is a PRO comprised of a single item rated on a scale from 0 ("No itch") to 10 ("Worst imaginable itch").
Study B: Proportion of participants with weekly average of daily WI-NRS <2 at Week 12 | Week 12
  WI-NRS is a PRO comprised of a single item rated on a scale from 0 ("No itch") to 10 ("Worst imaginable itch").
Study B: Absolute change from baseline in weekly average of daily itch-related sleep disturbance NRS at Week 12 and Week 24 | Baseline to Week 12 and Week 24
  The sleep disturbance NRS is to be used by the participants to report the degree of their sleep loss related to itch over the past 24 hours. Participants will rate their sleep disturbance from 0 ('no sleep loss related to itch') to 10 ('I cannot sleep at all due to itch') once daily in the morning.
Study B: Percent change from baseline in weekly average of daily itch-related sleep disturbance NRS at Week 12 and Week 24 | Baseline to Week 12 and Week 24
  The sleep disturbance NRS is to be used by the participants to report the degree of their sleep loss related to itch over the past 24 hours. Participants will rate their sleep disturbance from 0 ('no sleep loss related to itch') to 10 ('I cannot sleep at all due to itch') once daily in the morning.
Study B: Change from baseline in DLQI score at Week 12 and Week 24 | Baseline to Week 12 and Week 24
  The DLQI is a validated 10-item questionnaire to measure dermatology-specific quality of life (QoL) in adult patients. Overall scoring ranges from 0 to 30, with a higher score indicating a poorer QoL.
Study B: Change from baseline in the ItchyQoL score at Week 12 and Week 24 | Baseline to Week 12 and Week 24
  ItchyQoL is a pruritus-specific QoL instrument that measures specifically disease burden in pruritus patients. It is a 22-item instrument that measures the degree to which pruritus affects quality-of-life for the past week. The overall score is the average of the 22 items ranging from 1 to 5. A higher score corresponds to a more adverse impact on QoL.
Study B: Change from baseline in HADS total score at Week 12 and Week 24 | Baseline to Week 12 and Week 24
  The HADS is a validated questionnaire for screening anxiety and depression in non-psychiatric populations. The total score ranges from 0 to 42. 0 to 7= normal; 8 to 10= borderline abnormal; 11 to 21= abnormal.
Study B: Percentage of participants experiencing TEAEs or SAEs from baseline through EOS | Baseline to Week 36
  Percentage of participants experiencing TEAEs or SAEs from baseline through EOS
Study B: Incidence of treatment-emergent ADA against dupilumab | Baseline to Week 36
  Incidence of treatment-emergent ADA against dupilumab

CONTACTS AND LOCATIONS:
Locations (84):
- United States (18):
  - Kern Allergy and Medical Research- Site Number : 8400016, Bakersfield, California
  - Modena Allergy + Asthma- Site Number : 8400038, La Jolla, California
  - FoxHall Dermatology- Site Number : 8400042, Washington D.C., District of Columbia
  - Palm Harbor Dermatology- Site Number : 8400024, Belleair, Florida
  - University of Miami Hospital- Site Number : 8400011, Miami, Florida
  - Skin Care Physicians of Georgia - Macon- Site Number : 8400030, Macon, Georgia
  - Aeroallergy Research Laboratory- Site Number : 8400036, Savannah, Georgia
  - Dawes Fretzin Clinical Research- Site Number : 8400007, Indianapolis, Indiana
  - Dermatology Specialists Research (DS Research) - Kentucky- Site Number : 8400031, Louisville, Kentucky
  - Tulane University Health Sciences Center- Site Number : 8400045, New Orleans, Louisiana
  - Johns Hopkins Hospital- Site Number : 8400020, Baltimore, Maryland
  - The Asthma and Allergy Center- Site Number : 8400014, Bellevue, Nebraska
  - Icahn School of Medicine at Mount Sinai- Site Number : 8400034, New York, New York
  - AXIS Clinicals - Fargo- Site Number : 8400037, Fargo, North Dakota
  - Optima Research - Boardman- Site Number : 8400039, Boardman, Ohio
  - Columbia Dermatology & Aesthetics- Site Number : 8400047, Columbia, South Carolina
  - National Allergy and Asthma - North Charleston - Northside Drive- Site Number : 8400032, North Charleston, South Carolina
  - Complete Dermatology - Sugar Land- Site Number : 8400046, Sugar Land, Texas
- Argentina (8):
  - Investigational Site Number : 0320004, Rosario, Santa Fe Province
  - Investigational Site Number : 0320008, Rosario, Santa Fe Province
  - Investigational Site Number : 0320005, Buenos Aires
  - Investigational Site Number : 0320001, Buenos Aires
  - Investigational Site Number : 0320006, Buenos Aires
  - Investigational Site Number : 0320007, Buenos Aires
  - Investigational Site Number : 0320002, Buenos Aires
  - Investigational Site Number : 0320003, Buenos Aires
- Canada (7):
  - Investigational Site Number : 1240001, Calgary, Alberta
  - Investigational Site Number : 1240008, Edmonton, Alberta
  - Investigational Site Number : 1240002, London, Ontario
  - Investigational Site Number : 1240003, Markham, Ontario
  - Investigational Site Number : 1240006, Toronto, Ontario
  - Investigational Site Number : 1240005, Montreal, Quebec
  - Investigational Site Number : 1240004, Verdun, Quebec
- China (9):
  - Investigational Site Number : 1560003, Beijing
  - Investigational Site Number : 1560004, Chengdu
  - Investigational Site Number : 1560009, Chongqing
  - Investigational Site Number : 1560006, Guangzhou
  - Investigational Site Number : 1560005, Guangzhou
  - Investigational Site Number : 1560002, Hangzhou
  - Investigational Site Number : 1560001, Shanghai
  - Investigational Site Number : 1560011, Suzhou
  - Investigational Site Number : 1560008, Wuhan
- Germany (2):
  - Investigational Site Number : 2760002, Berlin
  - Investigational Site Number : 2760003, Mainz
- Hungary (5):
  - Investigational Site Number : 3480001, Budapest
  - Investigational Site Number : 3480009, Budapest
  - Investigational Site Number : 3480005, Debrecen
  - Investigational Site Number : 3480003, Szeged
  - Investigational Site Number : 3480002, Zalaegerszeg
- Italy (7):
  - Investigational Site Number : 3800004, Torette, Ancona
  - Investigational Site Number : 3800007, Cona, Ferrara
  - Investigational Site Number : 3800005, Florence, Firenze
  - Investigational Site Number : 3800003, Milan, Milano
  - Investigational Site Number : 3800002, Rozzano, Milano
  - Investigational Site Number : 3800006, Naples, Napoli
  - Investigational Site Number : 3800001, Rome, Roma
- Japan (7):
  - Investigational Site Number : 3920007, Urayasu, Chiba
  - Investigational Site Number : 3920003, Obihiro, Hokkaido
  - Investigational Site Number : 3920006, Sapporo, Hokkaido
  - Investigational Site Number : 3920004, Habikino, Osaka
  - Investigational Site Number : 3920002, Sakai, Osaka
  - Investigational Site Number : 3920005, Izumo, Shimane
  - Investigational Site Number : 3920001, Tachikawa, Tokyo
- Poland (5):
  - Investigational Site Number : 6160001, Krakow, Lesser Poland Voivodeship
  - Investigational Site Number : 6160007, Wroclaw, Lower Silesian Voivodeship
  - Investigational Site Number : 6160003, Wroclaw, Lower Silesian Voivodeship
  - Investigational Site Number : 6160008, Warsaw, Masovian Voivodeship
  - Investigational Site Number : 6160005, Warsaw, Masovian Voivodeship
- South Korea (7):
  - Investigational Site Number : 4100003, Busan, Busan
  - Investigational Site Number : 4100004, Ansan-si, Gyeonggi-do
  - Investigational Site Number : 4100005, Seoul, Seoul-teukbyeolsi
  - Investigational Site Number : 4100002, Seoul, Seoul-teukbyeolsi
  - Investigational Site Number : 4100006, Seoul, Seoul-teukbyeolsi
  - Investigational Site Number : 4100001, Seoul, Seoul-teukbyeolsi
  - Investigational Site Number : 4100007, Seoul, Seoul-teukbyeolsi
- Spain (5):
  - Investigational Site Number : 7240003, Barcelona, Barcelona [Barcelona]
  - Investigational Site Number : 7240006, Barcelona, Catalunya [Cataluña]
  - Investigational Site Number : 7240001, Pontevedra, Pontevedra [Pontevedra]
  - Investigational Site Number : 7240005, Alicante
  - Investigational Site Number : 7240004, Córdoba
- Taiwan (4):
  - Investigational Site Number : 1580003, Kaohsiung City
  - Investigational Site Number : 1580004, New Taipei City
  - Investigational Site Number : 1580001, Taipei
  - Investigational Site Number : 1580002, Taoyuan

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: EFC16973 Chronic Pruritus of Unknown Origin Website — https://www.chic-clinicaltrial.com/
- See also: EFC16973 Plain Language Results Summary — https://sanofi.trialsummaries.com/Study/StudyDetails?id=25259&tenant=MT_SNY_9011